CLINICAL TRIAL: NCT05250388
Title: The Effect of Arthroscopic Bankart Repair on Anterior-posterior Glenohumeral Translation and Shoulder Proprioception in Patients With Traumatic Anterior Shoulder Instability: a Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Catarina Malmberg (Other)
Collaborators: Køge Hospital (Unknown); Herlev og Gentofte Hospital (Unknown); Adeas Hospitaler (Unknown); Gildhøj Privathospital (Unknown)
Responsible Party: Sponsor-Investigator, Catarina Malmberg, MD, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Other Study IDs: H-21027799
Record Dates: First submitted 2022-01-31; First posted 2022-02-22 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Shoulder Dislocation
Keywords: Traumatic anterior shoulder instability; Shoulder dislocation; Glenohumeral instability; Glenohumeral biomechanics; Shoulder biomechanics; Glenohumeral translation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Patients aged 18-40 years with symptomatic unilateral traumatic anterior shoulder instability, following radiographically confirmed or manually reduced dislocation (first-time or recurrent), scheduled for arthroscopic Bankart repair, and with no pathology in the contralateral shoulder.
  The study is not interventional but observational, examining biomechanical and proprioceptive conditions in patients' unstable shoulders before and after the surgical procedure.
  Interventions: Procedure: Arthroscopic Bankart repair

INTERVENTIONS:
Procedure: Arthroscopic Bankart repair — Arthroscopic Bankart repair is a minimally invasive surgical procedure with the aim to reattach and tighten the detached labrum and ligaments within the shoulder joint.

SUMMARY:
The purpose of the study is to investigate biomechanical and proprioceptive conditions in patients with symptomatic traumatic anterior shoulder instability undergoing arthroscopic Bankart repair. To determine these, non-invasive and non-irradiating examination methods that have been proven valid and reliable will be used in a combination that has not been reported before. The objective is to determine whether the anatomical reconstruction affects biomechanical and proprioceptive measures in the traumatic unstable shoulder. The study will also investigate patient-reported and clinical outcomes.

The hypotheses are that the intervention improves biomechanical and proprioceptive conditions to the near-normal state, as measured after both 6 and 12 months. Further, hypotheses are that the intervention leads to improved patient-reported and clinical outcomes.

DETAILED DESCRIPTION:
• Aim: To investigate the effect of arthroscopic Bankart repair on shoulder biomechanics and proprioception, and increase understanding of traumatic anterior shoulder instability.

• Main research questions: A (biomechanics): Does arthroscopic Bankart repair have a stabilising effect on the anterior-posterior glenohumeral translation in patients with traumatic anterior shoulder instability? B (proprioception): Does arthroscopic Bankart repair improve neuromuscular control in patients with traumatic anterior shoulder instability?

• Objectives and hypotheses research question A: In patients with traumatic anterior shoulder instability undergoing arthroscopic Bankart repair, to investigate the anterior-posterior glenohumeral translation and the scapular rotations before and six and twelve months after surgery and whether the ranges are restored to the same as the non-injured contralateral shoulder.

Hypotheses:

* Arthroscopic Bankart repair results in a ≥2.5 mm decrease in anterior-posterior glenohumeral translation, remaining both six and twelve months after surgery.
* Arthroscopic Bankart repair reduces anterior-posterior glenohumeral translation to the same range as measured in the non-injured shoulder (±2.5 mm).
* Arthroscopic Bankart repair reduces superior-inferior glenohumeral translation significantly, as measured six and twelve months after surgery.
* Scapular rotations and tilt remain unchanged after arthroscopic Bankart repair.

  * Objectives and hypotheses research question B:

In patients with traumatic anterior shoulder instability undergoing arthroscopic Bankart repair, to investigate the neuromuscular control before and six and twelve months after surgery and whether the neuromuscular control is restored to the same level as the non-injured contralateral shoulder.

Hypotheses:

* Arthroscopic Bankart repair improves neuromuscular control, remaining both six and twelve months after surgery.
* Arthroscopic Bankart repair improves neuromuscular control to the same range as the non-injured shoulder.

  * Other objectives:

In patients with traumatic anterior shoulder instability undergoing arthroscopic Bankart repair:

1. To investigate patient-reported outcome measures (PROM) before and six and twelve months after surgery.
2. To determine the recurrence rates (radiographically confirmed or manually reduced dislocation) in the first twelve months after surgery.
3. To investigate the shoulder range of motion (ROM) before and six and twelve months after surgery.
4. To assess the joint instability by manual testing before and six and twelve months after surgery.
5. To quantify potential bone loss before surgery.
6. To investigate if there are correlations between a) the shoulder biomechanics and b) the neuromuscular control, and PROM, ROM, and bone loss, respectively.

   * Type of study:

Multi-clinical prospective cohort study including 30 patients. Patients' contralateral shoulders will be used as controls.

• Time schedule: Recruitment and inclusion began 1 April 2022 and is expected to last for 24 months. With a one-year follow-up the complete study period is expected to last three years.

* Set-up: Five sports orthopaedics clinics in the Capital Region of Denmark will recruit patients for the study. While the responsibility for treatment remains at the recruiting center, all study-related activities will take place at the Copenhagen University Hospital Hvidovre. Patients who have signed an informed consent form will undergo examinations prior to, as well as six and twelve months after surgery. All examinations will include biomechanical and proprioceptive testing, accompanied by a clinical shoulder examination and two validated electronic questionnaires regarding shoulder-related function and quality of life. A pre-interventional 3D computed tomography scan will be performed to evaluate bone loss. Study participation will not influence the treatment course.
* Sample size calculation:

The sample size calculation is made to allow for assessment of the primary outcomes within each category of outcomes; For research question A concerning biomechanics, the study is powered to detect a mean change in anterior-posterior glenohumeral translation of ≥2.5 mm with a standard deviation (SD) of 2.3 mm. For research question B concerning neuromuscular control, the study is powered to detect an effect size of 0.8 for change in reaction time. For the clinical and patient-reported outcomes, the study is powered to detect an effect size of 0.8 for the WOSI score.

For power of 90% and type I error rate of 0.017 (0.05/3), correcting for three tests, sample size for a one-sample t-test is 15, 24 and 24 for anterior-posterior glenohumeral translation, reaction time and WOSI score, respectively. As such, the largest sample size of 24 will be used. To account for expected dropout rate of 25% a total of 30 patients will be included.

Originally, the study was powered to detect a between group difference in anterior-posterior glenohumeral translation of ≥2.5 mm with a standard deviation (SD) of 2.3 mm, and a power of 80%. With six variables in the analysis (sex, height, BMI, dominant/non-dominant side affected, bone loss, clinical score) and an estimated 15% dropout rate, the calculation resulted in 55 patients. During the writing of a protocol article, it was realized that since the same shoulders are compared pre and post intervention no between groups analysis is performed and hence the setup controls for the six mentioned variables in itself. The sample size was thus re-calculated as stated above.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Unilateral traumatic anterior shoulder instability booked for arthroscopic Bankart repair according to the department's guidelines (extent of symptoms, suffer recurrent dislocations, positive apprehension and relocation test, limited bone loss)
* Willing to adhere to the study protocol, herein attend follow-up
* The patient must be able to speak and understand Danish
* The patient must be able to give written informed consent

Exclusion Criteria:

* Traumatic instability in the opposite shoulder
* For one or both shoulders: posterior, multi-directional or atraumatic instability
* For one or both shoulders: traumatic rotator cuff or biceps tendon tear, Superior Labrum from Anterior to Posterior tear (SLAP-lesion)
* For one or both shoulders: traumatic fracture of proximal humerus (other than Hill-Sachs lesion), clavicula, scapula (other than glenoid) or dislocation of sternoclavicular or acromioclavicular joints
* For one or both shoulders: atraumatic shoulder pathologies (e.g. frozen shoulder, symptomatic osteoarthritis of the shoulder or acromioclavicular joints, acute calcific tendinitis)
* Pregnancy
* Terminal illness or severe medical illness: American Society of Anesthesiology (ASA) score ≥3.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged 18-40 years with unilateral symptomatic traumatic anterior shoulder instability undergoing arthroscopic Bankart repair
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in anterior-posterior glenohumeral translation (range in millimeters) | baseline, 6 months
  The effect of Bankart repair on anterior-posterior glenohumeral translation, measured 6 months after intervention and compared to pre-interventional. The translation will be measured using ultrasound examination.

SECONDARY OUTCOMES:
Change in anterior-posterior glenohumeral translation (range in millimeters) | baseline, 12 months
  Longer-term effects of Bankart repair on anterior-posterior glenohumeral translation, as measured 12 months after intervention and compared to pre-interventional. The translation will be measured using ultrasound examination.
Change in neuromuscular control (as assessed with the Copenhagen Assessment of Neuromuscular Control in the Unstable Shoulder (CANCUS) protocol). | baseline, 6 months, 12 months
  The effect of Bankart repair on neuromuscular control at 6 and 12 months after intervention and compared to pre-interventional. Neuromuscular control will be assessed using the Copenhagen Assessment of Neuromuscular Control in the Unstable Shoulder (CANCUS) protocol.
Change in superior-inferior glenohumeral translation (range in millimeters) | baseline, 6 months, 12 months
  Effects of Bankart repair on superior-inferior glenohumeral translation, measured 6 and 12 months after intervention and compared to pre-interventional.
Change in scapular rotations (degrees) | baseline, 6 months, 12 months
  Effects of Bankart repair on scapular rotations, measured 6 and 12 months after intervention and compared to pre-interventional.

OTHER OUTCOMES:
Instability tests | baseline, 6 months, 12 months
  The effect of Bankart repair on clinical instability tests: sulcus sign, load and shift, apprehension test and relocation test.
Change in Western Ontario Shoulder Instability (WOSI) Index | baseline, 6 months, 12 months
  The Western Ontario Shoulder Instability (WOSI) Index is a patient-reported outcome measure (PROM).
  It consists of 21 items, each scored on a 100mm Visual Analogue Scale (VAS). Each item falls into one of the domains of physical function, sports/recreation/work, lifestyle and emotional well-being. Each question is scored between 0-100 points and the summation of all the questions results in a final WOSI score. The final score ranges from 0 (best possible score - the patient is experiencing no decrease in shoulder-related quality of life) to 2100 (worst score - signifies extreme distress in shoulder-related quality of life).
Change in EQ-5D(-5L) questionnaire on quality of life | baseline, 6 months, 12 months
  The EQ-5D-5L questionnaire on quality of life is a patient-reported outcome measure (PROM), with five components, which assess the severity of problems in three functional dimensions (mobility, self-care, and usual activities) and two somatic symptom dimensions (pain/discomfort and anxiety/depression). The response scales consist of a heading and five short statements, each describing a different level of severity within the dimensions.
Change in degrees of shoulder range of motion | baseline, 6 months, 12 months
  Range of motion will be assessed clinically as degrees from anatomical position in the following planes: flexion, extension, scaption, internal and external rotation.
Bone loss | baseline
  A pre-surgical computed tomography (CT) scan to measure potential bone loss. Glenoid bone loss is measured using the PICO-method, which is based on calculating the size of the defect as the percentage of a best-fit circle from the contralateral glenoid. The size (the largest height, width and depth in millimeters) of Hill-Sachs lesions on the humeral head is also measured and registered, but not the specific location.
Recurrent events | 6 months, 12 months
  Any radiographically confirmed or manually reduced dislocations in the first twelve months are registered during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Malmberg, MD, Principal Investigator — Dept. of Orthopedic Surgery, Copenhagen University Hospital Hvidovre
Locations (1):
- Dept. of Orthopedic Surgery, Copenhagen University Hospital Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malmberg C, Andreasen KR, Bencke J, Kjaer BH, Holmihc P, Barfod KW. Reliability of ultrasound measurement of glenohumeral instability. Dan Med J. 2025 Oct 15;72(11):A11240835. doi: 10.61409/A11240835. PMID 41133330
- [Derived] Malmberg C, Andreasen KR, Bencke J, Kjaer BH, Holmich P, Barfod KW. Biomechanical and neuromuscular characteristics in patients with traumatic anterior shoulder instability undergoing arthroscopic Bankart repair: a clinical prospective cohort study protocol. BMJ Open. 2024 Mar 1;14(3):e078376. doi: 10.1136/bmjopen-2023-078376. PMID 38431300